CLINICAL TRIAL: NCT06634992
Title: Paediatric Observatory of Oral Food Tolerance Induction in the Allergy Department of the Saint-Vincent de Paul Hospital in Lille
Brief Title: Observatory of the Lille Paediatric Allergy Unit
Acronym: PAUL
Status: Recruiting | Type: Observational
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Other Study IDs: RNIPH-2021-36
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Child Allergy; IgE-Mediated Allergic Process; Food Allergy
Keywords: Food allergy; Food challenge test; IgE-Mediated; Observatory
MeSH Terms: conditions — Food Hypersensitivity | interventions — Immunotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Allergy to hazelnut, walnut, pistachio, cashew or peanut
  Interventions: Other: Oral immunotherapy
- Group 2: Allergy to cow's milk, wheat or egg
  Interventions: Other: Oral immunotherapy
- Group 3: Allergy to unusual foods: sesame, celery, fenugreek, peas, lentils or others
  Interventions: Other: Oral immunotherapy

INTERVENTIONS:
Other: Oral immunotherapy — Clinical Follow up

SUMMARY:
The goal of this study is to set up a paediatric observatory within the allergology department of The saint Vincent Hospital, Lille. The study aims to:

• Collect exhaustive prospective data from patients eligible for oral immunotherapy.

This prospective observatory will enable statistical analyses to be carried out on common food allergens such as hazelnut, cashew nut, pistachio and others.

DETAILED DESCRIPTION:
During the consultation, the allergist will inform the legal representative and the child about the terms of the study, and will provide them with an information note specifying the objectives of the study and its terms, the involvement of the child and his or her rights.

Depending on the allergen involved, the oral immunotherapy session will be assigned to one of three study groups: 1) allergen to hazelnut, walnut, pistachio, cashew or peanut,2) allergen to cow's milk, wheat or egg, 3) allergen to unusual foods: sesame, celery, fenugreek, peas, lentils, etc.

For each patient, and for each visit during the treatment period the collection of anthropometric, sociodemographic and medical data relating to oral food challenge will be done

Oral immunotherapy will then be started in accordance with standard practice. During this first visit, the investigator will give the patient a diary in which to record information about any IgE-mediated side-effects of the oral immunotherapy. Subsequent visits will follow the patient's usual routine until the desensitisation threshold is reached or the patient decides to stop the oral immunotherapy protocol. Visits will be made every 6 months, with a window of two months around each date.During these monitoring visits, tthe collection of anthropometric, sociodemographic and medical data relating to oral food challenge will be continue.

During each visit, a new food challenge test may be performed at the investigator's discretion to assess a new reactogenic threshold. Following this test, the following data will be collected:

* the cumulative dose ingested (mg food and mg food protein)
* the grade of the reaction (from 0 to 5 according to the Astier et Coll classification)
* achievement of desensitisation

A patient begins oral immunotherapy following food challenge test in a day hospital. Thus, a patient consulting at different times for several allergies and eligible for several oral immunotherapies will be able to take part in the study for several allergens. The follow-up of the different oral immunotherapies started (maximum 2 simultaneously, but could go up to 5, 6... over time) will be distinct. The patient may therefore participate several times in the study: in different groups, or in the same group, for different allergens. All the above data are collected separately for each new oral immunotherapy (except for socio-demographic data and information on previous oral immunotherapies, which are collected only at the time of inclusion).

In very rare cases, a patient may undergo several oral immunotherapies for the same allergen, but only the first oral immunotherapy (from the time the observatory was set up) will be taken into account in this study. If oral immunotherapy for the same allergen has already been carried out before the observatory was set up, the second oral immunotherapy for this allergen will not be included in the study, as its results will be biased.

ELIGIBILITY:
Inclusion criteria:

* patient under 15 years and 9 months,
* positive diagnosis of food allergy (positive food challenge test or "highly probable allergy", defined by a convincing history, a positive prick test and IgE > 0.35 kUA/L),
* eligible for oral food challenge
* accepting the following allergens : hazelnut, walnut, pistachio, cashew, peanut, cow's milk, wheat, egg, sesame, celery, fenugreek, pea, lentils or others

Exclusion criteria:

* Opposition
* Already received oral challenge for the same allergen.

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All eligible patients consulting at the allergology service of the Saint Vincent Hospital, Lille, France will be informed and included, unless they object.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Age | at inclusion
  For each patient, and for each visit during the treatment period the collection of anthropometric, sociodemographic and medical data relating to oral food challenge will be done
Sex | at inclusion
  For each patient, and for each visit during the treatment period the collection of anthropometric, sociodemographic and medical data relating to oral food challenge will be done
Oral immunotherapies followed before inclusion | at inclusion
  For each patient, and for each visit during the treatment period the collection of anthropometric, sociodemographic and medical data relating to oral food challenge will be done
Determination of comorbidities | at inclusion
  For each patient, and for each visit during the treatment period the collection of anthropometric, sociodemographic and medical data relating to oral food challenge will be done
Determination of allergen under consideration | at inclusion
  For each patient, and for each visit during the treatment period the collection of anthropometric, sociodemographic and medical data relating to oral food challenge will be done
Specific IgE | at inclusion
  For each patient, and for each visit during the treatment period the collection of anthropometric, sociodemographic and medical data relating to oral food challenge will be done
Recombinants | 5 years
  For each patient, and for each visit during the treatment period the collection of anthropometric, sociodemographic and medical data relating to oral food challenge will be done
Cumulative ingested dose | 5 years
  This dose will be determined by mg/food and m/ food protein
Allergic reaction according to the Astier and Coll classification | 5 years
  Astier score for anaphylaxis according to symptoms:
  0- Absent
  1- Abdominal pain spontaneous resolution, Urticaria < 10 papules, Eczema, Rhinoconjunctivitis 2-1 Organ affected, Abdominal pain requiring treatment, Angioedema with laryngeal involvement, Moderate asthma: cough and PEF > 20%.
  3- 2 Affected organs 4- 3 organs affected or Asthma attack requiring treatment or Laryngeal edema or Arterial hypotension 5- Cardiorespiratory impairment requiring ICU admission
Type of oral challenge | 5 years
  Type of ingested food during the oral immunotherapy: fresh food / industrial products
Reception of emergency kit | 5 years
  If the reception of an emergency kit was needed will be determined by yes/no
Second oral food challenge | 5 years
  If a second oral challenge was needed will be determined by yes/no
Tolerance according to reactogenic thresholds for allergens | 5 years
  Subsequent visits will follow the patient's usual routine until the desensitisation threshold is reached or the patient decides to stop the oral immunotherapy protocol.
Amount of reactions IgE mediated | 5 years
  Subsequent visits will follow the patient's usual routine until the desensitisation threshold is reached or the patient decides to stop the oral immunotherapy protocol.
Amount of reactions non IgE mediated | 5 years
  Subsequent visits will follow the patient's usual routine until the desensitisation threshold is reached or the patient decides to stop the oral immunotherapy protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Tomas MORALY, Principal Investigator — Groupement des Hopitaux de l'institut catholique de Lille
Locations (1):
- Groupement de l'Institut Catholique de Lille - Hôpital Saint Vincent de Paul, Lille, France

IPD SHARING:
Plan to Share IPD: No